CLINICAL TRIAL: NCT00890513
Title: Family Satisfaction in the Intensive Care Unit - a Multicentre Assessment
Acronym: Swiss-BEAN
Status: Completed | Type: Observational
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Rothen Hans Ulrich, Department of Intensive Care Medicine, University Hospital Bern, Switzerland
Other Study IDs: KEK_180/06
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2009-11-20 (Estimated); Status verified 2009-11

CONDITIONS: Critical Illness
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The primary aim of the present study is to assess satisfaction in a large sample of next of kin in Swiss-German ICUs.

Secondary aims are to test the hypothesis that family satisfaction is related to ICU structure and process and to factors related to patients and next of kin. Further, the hypothesis will be tested that proxy assessment is possible, i.e. next of kin rate satisfaction with care similar to patients.

ELIGIBILITY:
Inclusion Criteria:

* family members of patients staying for > 48 hours in an ICU

Exclusion Criteria:

* lack of consent,
* insufficient knowledge of German language

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Next of kin of patients cared for in one of the 42 ICU's located in german-speaking Switzerland (ICU recognized by Swiss Society of Intensive Care Medicine).
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2007-04; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To assess satisfaction in Swiss-German ICUs

SECONDARY OUTCOMES:
To test the hypothesis that family satisfaction is related to ICU structure and process To test the hypothesis that proxy assessment is possible

CONTACTS AND LOCATIONS:
Overall Officials: Hans U Rothen, MD PhD, Principal Investigator — Bern University Hospital, University of Bern-Switzerland
Locations (1):
- Department of Intenisve Care Medicine, Inselspital, Bern, Canton of Bern, Switzerland

REFERENCES:
- [Result] Stricker KH, Kimberger O, Schmidlin K, Zwahlen M, Mohr U, Rothen HU. Family satisfaction in the intensive care unit: what makes the difference? Intensive Care Med. 2009 Dec;35(12):2051-9. doi: 10.1007/s00134-009-1611-4. PMID 19730813
- [Derived] Stricker KH, Kimberger O, Brunner L, Rothen HU. Patient satisfaction with care in the intensive care unit: can we rely on proxies? Acta Anaesthesiol Scand. 2011 Feb;55(2):149-56. doi: 10.1111/j.1399-6576.2010.02293.x. Epub 2010 Sep 6. PMID 20825369